CLINICAL TRIAL: NCT00542646
Title: Pilot Study to Evaluate the Safety and Preliminary Efficacy of the Peritec Peritoneal Lined Stent and Delivery System
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PeriTec Biosciences Ltd. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PB-PLS-2005-001
Record Dates: First submitted 2007-10-10; First posted 2007-10-11 (Estimated); Last update posted 2007-11-28 (Estimated); Status verified 2007-11

CONDITIONS: Vascular Disease, Peripheral
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Endovascular Intervention — Peritoneal Lined Stent Endovascular Intervention

SUMMARY:
The occurrence of Peripheral Vascular Disease has been increasing which includes the large artery in the upper leg called Superficial Femoral Artery (SFA). The Peritoneal Lined Stent has been developed as a new method for treating narrowed area in the SFA. This research study will determine the safety and effectiveness of the Peritoneal Lined Stent in keeping th Superficial Femoral Artery open and allowing blood to flow in the leg.

ELIGIBILITY:
Inclusion Criteria:

* Patient with claudication or ischemic rest pain(Rutherford Categories 2-4)
* The angiogram will need to have been performed confirming superficial femoral artery short segment occlusion(<5cm first two patients and <10cm there on) or high grade(>50%)stenosis
* Patient has a signed and dated informed consent
* Patient has a resting ABI <0.9 or an abnormal exercise ABI if resting ABI is normal. Patients with incompressible arteries (ABI >1.2) must have TBI <0.8
* Life expectancy greater than one year
* The ability to comply with protocol follow up requirements and required testing
* Angiographic lesion requirements assessed at time of procedure

  * Lesion of the superficial femoral artery with a short segment occlusion(<5cm first two patients and <10cm there on) or high grade (>50%) stenosis
  * Target lesion 1 cm below profunda/superficial femoral artery origin and 3cm above knee joint
  * Angiographic evidence of a minimum of at least one tibial with continuous artery runoff to the ankle that does not require intervention
  * Guidewire has successfully traversed lesion and is within the true lumen of the distal vessel, and successful placement of 9 french(Fr) sheath

Exclusion Criteria:

* Untreated iliac artery in-flow limiting lesion
* Significant proximal common femoral or superficial femoral artery disease above or below target lesion
* Any previously treated superficial femoral artery lesion
* Any previous stenting or surgery in the target vessel
* Femoral or popliteal aneurysm
* Non-Atherosclerotic disease resulting in occlusion (e.g. embolism, vasculitis,etc)
* Serum creatinine >2.5 mg/dl
* Any previously known coagulation disorder, including hypercoagulability
* Severe medical co-morbidities or other medical condition (for example untreated coronary heart disease and congestive heart failure, severe chronic obstructive pulmonary disease, metastasis malignance, etc.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2006-11; Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
Efficacy: Primary patency postprocedure and technical success Safety: Composite of major procedural adverse events | 30 Days

SECONDARY OUTCOMES:
Primary Patency Primary Assisted Patency Secondary Patency Clinical Success Major Amputations Target Vessel Revascularization Target Lesion Revascularization | 3 Months Intervals except for Target Lesion Revascularization at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Timur Sarac, MD, Study Director — PeriTec Bioscience Ltd
Locations (1):
- Pontificia Universidad Catolica de Chile, Santiago, Chile

REFERENCES:
- [Background] Carnevale K, Ouriel K, Gabriel Y, Clair D, Bena JF, Silva MB, Sarac TP. Biological coating for arterial stents: the next evolutionary change in stents. J Endovasc Ther. 2006 Apr;13(2):164-74. doi: 10.1583/05-1710R.1. PMID 16643070
- [Background] Sarac TP, Carnevale K, Smedira N, Tanquilut E, Augustinos P, Patel A, Naska T, Clair D, Ouriel K. In vivo and mechanical properties of peritoneum/fascia as a novel arterial substitute. J Vasc Surg. 2005 Mar;41(3):490-7. doi: 10.1016/j.jvs.2004.11.033. PMID 15838485